CLINICAL TRIAL: NCT05327231
Title: A Phase I, Open-label Clinical Trial to Evaluate Safety, Tolerability, Antitumor Activities and Pharmacokinetics of IN10018 as Mono or Combination Therapy in Locally Advanced or Metastatic Gastric or Gastroesophageal Junction Adenocarcinoma
Brief Title: IN10018 Monotherapy or in Combination With Docetaxel in Gastric or GEJ Adenocarcinoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: InxMed (Shanghai) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IN10018-003
Record Dates: First submitted 2022-03-29; First posted 2022-04-14 (Actual); Last update posted 2022-11-16 (Actual); Status verified 2022-09

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — Docetaxel

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- IN10018 Monotherapy (Experimental): Participants will be instructed to take IN10018 orally once daily at approximately the same time each day, to ensure a dose interval of approximately 24 hours.
  Interventions: Drug: IN10018
- IN10018 Combination with Docetaxel (Experimental): Participants will be instructed to take IN10018 orally once daily at approximately the same time each day, to ensure a dose interval of approximately 24 hours. Docetaxel 75mg/m2 every 21 days a cycle.
  Interventions: Drug: IN10018; Drug: Docetaxel

INTERVENTIONS:
Drug: IN10018 — IN10018 orally once daily at approximately the same time each day, to ensure a dose interval of approximately 24 hours.
Drug: Docetaxel — Docetaxel 75mg/m2 every 21 days a cycle.
  Arms: IN10018 Combination with Docetaxel

SUMMARY:
This is a phase I, multi-center clinical trial to evaluate the safety, tolerability, antitumor activities and pharmacokinetics of IN10018 as monotherapy or in combination with docetaxel in previously-treated locally advanced or metastatic gastric or gastroesophageal junction (GEJ) adenocarcinoma.

DETAILED DESCRIPTION:
Eligibility patients will be enrolled into the study and assigned to treatment groups: 1) IN10018 monotherapy group, and 2) IN10018+Docetaxel combination group. This study contains 2 parts of dose escalation and dose expansion for each treatment group. The monotherapy group will enroll patients failed to respond to standard therapy or standard or curative therapy does not exist or is not tolerable, and explore IN10018 monotherapy RP2D with the starting dose of IN10018 100mg QD per 3+3 design. The combination group will enroll patients who have disease progression within 3 months after at least first-line therapy, and explore IN10018+docetaxel RP2D with the starting dose of IN10018 100mg QD + docetaxel 75mg/m2 per 3+3 design. The dose expansion part will start after attaining the RP2D of IN10018 monotherapy and IN10018+docetaxel combination therapy.

ELIGIBILITY:
Inclusion Criteria:

* 1.Has histologically or cytologically confirmed diagnosis of locally advanced and/or metastatic gastric or GEJ adenocarcinoma.

  * For monotherapy, participants need to be failed to respond to standard therapy or standard or curative therapy does not exist or is not tolerable.
  * For combination therapy, participants need to have disease progression within 3 months after at least first-line therapy.
* 2.Has at least one measurable tumor lesion per RECIST 1.1.
* 3.Has an ECOG performance status of 0 or 1.
* 4.Estimated life expectancy is more than 3 months.
* 5.Adequate organ and bone marrow functions.
* 6.Has been fully informed and provided written informed consent for the study

Exclusion Criteria:

* 1.Has other histological types other than adenocarcinoma.
* 2.For participants with HER2/neu positive tumors or have an unknown tumor status, need to match the following:

  * If HER2/neu positive, participant must have documentation of disease progression on trastuzumab or other anti-HER2/neu therapy.
  * Participants with unknown status must have their HER2/neu status determined locally. If HER2/neu-negative, the participant will be eligible. If HER2/neu-positive, the participant must have documentation of disease progression on trastuzumab or other anti-HER2/neu therapy.
* 3.Has had disease progression after docetaxel/paclitaxel containing treatment (combination therapy only).
* 4.Has received prior systemic therapies (i.e. chemotherapy, biotherapy, endocrinotherapy, and immunotherapy) within 4 weeks prior to start of study treatment.
* 5.Has received prior radiotherapy within 2 weeks prior to start of study treatment.
* 6.Has severe allergy or hypersensitivity to IN10018 and/or docetaxel, or any components used in their preparation or has contraindication for taxane therapy. For participants in monotherapy group, only restriction to IN10018 applies.
* 7.Has severe renal disease or impaired renal function.
* 8.Has an active infection requiring systemic therapy within 2 weeks prior to start of study treatment.
* 9.Has a history or current evidence of interstitial lung disease.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2020-07-09 (Actual); Primary Completion 2021-12-03 (Actual); Study Completion 2022-03-31 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability in combination group | up to 24 months
  Number of patients with adverse event in combination group; Number of patients with laboratory abnormalities, abnormal vital signs and abnormal 12-lead ECG in combination group
DLTs in combination group | 21 days
  Number of patients with dose-limited toxicities (DLTs) in combination group
Phase II dose of IN10018 in combination with Docetaxel | up to 24 months
  Determine the recommended phase II dose (RP2D) of IN10018 in combination with Docetaxel

SECONDARY OUTCOMES:
Safety and tolerability in IN10018 monotherapy group | up to 24 months
  Number of patients with adverse event in monotherapy group; Number of patients with laboratory abnormalities, abnormal vital signs and abnormal 12-lead ECG in monotherapy group
DLTs in IN10018 monotherapy group | up to 24 months
  Number of patients with dose-limited toxicities (DLTs) in monotherapy group
Objective response rate (ORR) per RECIST v1.1 | up to 24 months
  Defined as the proportion of patients with complete response (CR) or partial response (PR).
Duration of objective response (DOR) per RECIST v1.1. | up to 24 months
  Defined as the time from start of the first documentation of CR or PR to the first documentation of disease progression or to death due to any cause, whichever comes first
Disease Control Rate (DCR) per RECIST v1.1. | up to 24 months
  Defined as the proportion of patients with CR, PR, or stable disease (SD)
Progression-free survival (PFS) per RECIST v1.1. | up to 24 months
  Defined as the time from start of study treatment to first documentation of disease progression or to death due to any cause, whichever comes first.
Overall survival (OS). | up to 30 months
  Defined as the time from the start of any study treatment to the date of death due to any cause.
Pharmacokinetics (PK):AUC | up to 24 months
  Area under the concentration-time curve (AUC).
Pharmacokinetics (PK):Cmax | up to 24 months
  PK: Maximum concentration (Cmax).
PK:Tmax | up to 24 months
  Time to Cmax (Tmax).
PK:Ctrough | up to 24 months
  Trough concentration (Ctrough).
PK:t1/2 | up to 24 months
  Elimination half-life (t1/2).
PK:CL/F | up to 24 months
  apparent clearance (CL/F).
PK:Vd/F | up to 24 months
  Apparent volume of distribution (Vd/F).

CONTACTS AND LOCATIONS:
Overall Officials: Jin Li, Doctor, Principal Investigator — Shanghai East Hospital
Locations (8):
- China (8):
  - Anyang Tumor Hospital, Anyang, Henan
  - Henan Cancer Hospital, Zhengzhou, Henan
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - The Affiliated Hospital of Nanjing University Medical School, Nanjing, Jiangsu
  - The First Hospital of China Medical University, Shenyang, Liaoning
  - Shanghai East Hospital, Shanghai, Shanghai Municipality
  - The First Affiliated Hospital of XI 'AN Jiaotong University, Xi’an, Shanxi
  - Tianjin Medical University Cancer Institute & Hospital, Tianjin, Tianjin Municipality